CLINICAL TRIAL: NCT04885504
Title: Post COVID-19 Biorepository
Status: Recruiting | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Leslie Spikes, MD, Associate Professor of Medicine, University of Kansas Medical Center
Other Study IDs: STUDY#00146337
Record Dates: First submitted 2021-05-11; First posted 2021-05-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Future projects might include genetic testing. Your sample may be sent to a lab for genetic testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Establish a biorepository, clinical data registry, and radiographic image database from individuals who were COVID positive at one time and are being seen for outpatient follow-up or a separate study visit.

DETAILED DESCRIPTION:
Living patients or their healthcare surrogates will provide informed consent prior to participation in the biorepository. Surrogate decision makers who cannot consent in person will be consented in accordance to the KUMC remote consent guidelines. Biospecimens to be collected include serum, plasma and whole blood. Blood samples will be collected during face-to-face encounters in the Post-COVID-19 clinic within the TUKHS pulmonary clinic or will be coordinated with other outpatient follow-up appointments (including separate procedure/lab-related visits) or separate study visits for ongoing, indepent studies. Samples will be collected at time of consent as well as at potential follow-up visits at approximately 3, 6, 12, and 12 months from enrollment. Blood samples will be processed, aliquoted, and stored at -80°C. A portion of the blood samples will be kept for DNA and RNA isolation, and a portion of plasma collected might be utilized to isolate peripheral blood mononuclear cells. Biospecimens will be labeled with the patient's study ID number, date of sample processing, and specimen type. Biospecimens will be stored through the duration of the study. If the patient chooses to withdraw consent, his or her samples in the biorepository will be destroyed. Biospecimens that have been previously used or disseminated will continue to be utilized. Future research may include whole genome testing, and these results will not be shared with the patient or their standard of care physician.

Patient data and historical radiographic imaging from after the date of consent will be collected using TUKHS medical records and stored in RedCap. The data to be collected is outlined in the data collection sheets.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is a patient at TUKHS or has agreed to participate in a study approved by the KUMC Human Research Protection Program (HRPP).
2. The participant has a previous diagnosis of COVID-19 confirmed by COVID-19 PCR or antibody testing and is being seen for outpatient follow-up.
3. Patient is ≥ 18 years of age or older.

Exclusion Criteria:

1. Participant declines to participate.
2. Participant or healthcare surrogate is unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participant will be recruited from the population of recovering COVID-19 patients seen in the Post-COVID-19 clinic within the TUKHS pulmonary clinic or who are scheduled for other outpatient appointments or unrelated study visits for separate, ongoing studies at TUKHS.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Establish a Biorepository | From Enrollment to 24 Months
  Establish a collection of biospecimens from patients who have recovered from COVID-19.
Develop Connections in Relation to Post-COVID Infection | From Enrollment to 12 Months
  Establish links between biospecimens, individual patient data and radiographic imaging, which will be collected and stored in RedCap.
Develop of Patient Registry | From Months 12 to 36
  Provide biospecimens and unique patient data to researchers investigating COVID-19 and its recovery. Separate IRB approval will be required for these studies.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Spikes, MD, Principal Investigator — University of Kansas Medical Center; Luigi R Boccardi, Ed.D., MPH, Study Director — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
The plan will be discussed between the Principal Investigator and the PI requesting access to Biospecimens.
Supporting Information: Study Protocol, ICF, CSR